CLINICAL TRIAL: NCT02723851
Title: An Open Label Study for Determining the Optimal Cut-off Point of Peak Endocardial Acceleration Measured by Corsens Device for Discriminating Between MI and Non-MI Subjects
Brief Title: Determining the Optimal Cut-off Point of PEA by Corsens Device for Discriminating Between MI and Non-MI Subjects
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Corsens Medical LTD (Industry)
Responsible Party: Sponsor
Other Study IDs: CS-COP-1
Record Dates: First submitted 2016-03-17; First posted 2016-03-31 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Acute MI patients: Corsens Recording and calculating Peak Endocardial Acceleration (PEA) Myocardial Contractility Index [MCI] and isovolumetric contraction (IVCT).
  Interventions: Device: Corsens
- Non-MI patients: Corsens Recording and calculating Peak Endocardial Acceleration (PEA) Myocardial Contractility Index [MCI] and isovolumetric contraction (IVCT).
  Interventions: Device: Corsens

INTERVENTIONS:
Device: Corsens — Recording and calculating Peak Endocardial Acceleration (PEA) Myocardial Contractility Index [MCI] and isovolumetric contraction (IVCT). Measurements will not affect the treatment provided to the patients.

SUMMARY:
Acute Myocardial Infarction (MI) is still the leading cause of death in the western world. Early warning (chest pain) signs of an acute MI are often misinterpreted and disregarded. In average it takes between 2-3 hours from the beginning of the chest pain. The damage to the heart in these 2 hours is critical and often irreversible. Thus an early warning test or device is highly warranted.

Corsens has developed a noninvasive device using several sensors applied to the chest and a detection system able to recognize the ischemic origin of chest pain. This clinical study is intended for evaluating the safety and efficacy of the Corsens technology while use for myocardial infarction detection

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the cardiac care unit (CCU) with ST elevation acute MI (STEMI) within 4 hours from beginning of chest pain.
* Male or female subjects aged 18 years or more (with no upper limit), of any race.
* Subjects willing to participate as evidenced by signing the written informed consent.

Exclusion Criteria:

* Obese patients with BMI>35.
* Subjects with cardiac arrhythmias including atrial fibrillation. Previous MI.
* Patients after coronary artery bypass grafting
* Unstable hemodynamic condition.
* Patient that can't or do not wish to sign the Inform Consent Form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with ST-elevation acute MI will be recruited to the study. Additional data that was already recorded in previous study from non-MI patients hospitalized for routine elective catheterization will be used.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-03 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0" to verify safety | 1 day
  To verify the safety of the Corsens technology while use for myocardial infarction detection.

SECONDARY OUTCOMES:
To define the optimal cut-off point (in terms of sensitivity and specificity) of the PEA measured by Corsens technology for discriminating between MI and non-MI patient. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Eugenia Nikolsky, Prof., Principal Investigator — Rambam Medical Center, Haifa Israel

IPD SHARING:
Plan to Share IPD: No